CLINICAL TRIAL: NCT04355286
Title: Ultraviolet Filter Bemotrizinol (BEMT): Clinical Pharmacokinetics Evaluation in a Topical Maximum Usage Trial (MUsT)
Brief Title: Bemotrizinol UV Filter Part 1 Clinical PK Evaluation in Topical MUsT Study
Acronym: BEMT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEMT-001
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Absorption; Chemicals; Sunscreening Agents
MeSH Terms: interventions — bis-ethylhexyloxyphenol methoxyphenyl triazine

STUDY DESIGN:
Intervention Model Description: Part 1 is an open label, 1-arm pilot study to evaluate the effects of multiple applications of a topical sunscreen formulation in healthy adult subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1, one-arm open label pilot study (Experimental): Part 1 is an open label, 1-arm pilot study to evaluate the systemic absorption and effects of multiple applications of a market-image topical sunscreen formulation containing BEMT (6%) under maximum use conditions in healthy adult subjects.
  Interventions: Drug: Bemotrizinol

INTERVENTIONS:
Drug: Bemotrizinol — Market-image topical sunscreen formulation containing BEMT (6%)
  Other Names: Bis-ethylhexyloxyphenol Methoxyphenyl Triazine, BEMT, PARSOL Shield, Tinosorb S, UNII-PWZ1720CBH, CAS: 187393-00-6

SUMMARY:
This will be a single clinical study conducted in 2 parts (Part 1: pilot study and Part 2: pivotal study).

Part 1 is an open-label, 1-arm study in 14 healthy adult subjects with the following primary objectives:

* Primary: To explore whether the active component, bemotrizinol (BEMT), is absorbed from a high-penetrating sunscreen formulation including 6% BEMT into the systemic circulation when applied under maximal-use conditions.
* Secondary: To obtain information needed for a successful pivotal study such as preliminary pharmacokinetic (PK) data, validation of study and analytical procedures, and the number of subjects needed.

Part 2 is an open-label, randomized, 3-arm study in 42 healthy adult subjects with the following objective:

• Primary: To assess the systemic absorption and pharmacokinetics of BEMT from 3 market image sunscreen formulations under maximal-use conditions.

DETAILED DESCRIPTION:
This will be a single clinical study conducted in 2 parts (Part 1: pilot study and Part 2: pivotal study). The duration of study participation will be approximately 42 days for Part 1, including a 30-day screening period, a 4-day treatment period (Days 1-4), and subjects leaving the clinical research unit (CRU) on the morning of Day 5. Subjects will then return to the CRU for follow-up visits on Days 8 and 12. On Day 12, End-of-Study activities will be completed. For Part 2, the duration of participation will be approximately the same, 42 days, and may be adjusted based on the results of Part 1.

Part 1 is an open-label, 1-arm pilot study to evaluate the effects of multiple applications of a topical sunscreen formulation in healthy adult subjects. It will include 14 subjects (7 male and 7 female) that will be admitted to the CRU on Day -1.

On the morning of Days 1 through 4, subjects will receive a topical application of the study drug between 07:00 and 10:00 hours followed by 3 more applications each day at 2, 4, and 6 hours after the first application, resulting in study drug application at 0, 2, 4, 6, 24, 26, 28, 30, 48, 50, 52, 54, 72, 74, 76, and 78 hours relative to the first application. The weight of study drug will be measured and recorded before and after dosing for each subject and each dose will be applied by a qualified person from the CRU.

Blood samples will be collected for the determination of plasma concentrations of BEMT from before the first topical application of study drug to 264 hours after the first study drug application.

Part 2 is an open-label, randomized, 3-arm pivotal study to evaluate the pharmacokinetics of BEMT after multiple applications of a topical sunscreen formulation in healthy adult subjects and may be modified based on observations from Part 1 and the Food and Drug Administration (FDA) revision. Part 2 will include 14 subjects (7 male and 7 female) in each arm. At least 3 formulations will be selected based on the plasma exposure data from the pilot study (Part 1), the in vitro permeation testing (IVPT) results, and the market survey for BEMT-containing formulations. All 42 subjects will be admitted to the CRU on Day -1 and randomly assigned to a treatment arm before study drug application on Day 1.

On the morning of Day 1, the assigned study drug will be applied topically between 07:00 and 10:00 hours; on Days 2, 3, and 4, subjects will receive an initial application at the same time as on Day 1 and 3 more topical applications at 2, 4, and 6 hours after the first application, resulting in study drug application at 0, 24, 26, 28, 30, 48, 50, 52, 54, 72, 74, 76, and 78 hours relative to the first application. The weight of study drug will be measured and recorded both before and after dosing for each subject and each dose will be applied by a qualified person from the CRU.

The PK blood sample collection schedule for Part 2 will be based on the results from Part 1. If significant systemic exposure is observed in Part 1, additional PK blood samples may be collected in Part 2 for assessment of metabolites.

In both parts of the study, In Parts 1 and 2, approximately 2 mg of active sunscreen ingredient per 1 cm2 of body surface area (calculation per method of Du Bois and Du Bois [1989]) will be evenly applied 4 times per study day (except for a 1-time application on the first day in Part 2) to areas of the body typically exposed to the sun: face (except eye area), ears, neck, torso, arms, and legs (at least 75% of the body surface area). The antecubital areas will be avoided and protected with an occlusive, self-adhesive cover when applying the sunscreen due to potential contamination of the sites used for PK blood sample collection. The topical applications of study drug will be administered with subjects in swim wear to simulate real world settings as well as for easy application. In addition to swim wear, subjects may wear scrubs in between applications and at other times throughout the day/night. Subjects are required to shower each morning after the first PK blood sample collection (and before the first application of the day), but not at other times during the day.

Safety evaluations will include adverse event (AE) monitoring, vital sign measurements, and physical examinations. All AEs reported by the subject or observed by the investigator or CRU staff will be recorded. Any AE reported after the informed consent form is signed and before study drug application will be recorded as medical history.

In the context of the Coronavirus (COVID-19) pandemic, the clinical site will follow all FDA, Centers for Disease Control and Prevention (CDC), and institutional review board (IRB) recommendations in its oversight and conduct of the trial. This may include changing the schedule of follow-up visits if it is considered necessary after a full risk/benefit analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following inclusion criteria will be eligible to participate in the study:

  1. Subject signs an IRB-approved written informed consent form (ICF) and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization) before any study-related procedures are performed.
  2. Subject is a healthy man or woman, 18 to 75 years of age, inclusive, who has a body mass index of 18.5 to 29.9 kg/m2, inclusive, at Screening.
  3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
  4. Subject has a negative test result for alcohol and drugs of abuse at Screening and Check-in (Day -1).
  5. Female subject is surgically sterile (hysterectomy, bilateral salpingo-oophorectomy, bilateral tubal ligation) or has a negative serum pregnancy test result before entry into the study and practices an adequate method of birth control (e.g., oral or parenteral contraceptives, hormonal or nonhormonal intrauterine device, barrier, abstinence) during the study and until 90 days after the last application of study drug.
  6. Male subject agrees to refrain from sexual activity with female partners unless an acceptable method of birth control is used by both partners. Male subject is surgically sterile or agrees to use barrier contraception (condom with spermicide), and refrain from sperm donation, from the first application of study drug until 90 days after the last application of study drug.
  7. Subject has a negative SARS-CoV-2 test result (polymerase chain reaction [PCR] method).
  8. Subject is highly likely (as determined by the investigator) to comply with the protocol-defined procedures and to complete the study.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be eligible to participate in the study:

  1. Subject who participated in Part 1 of the present maximum usage trial (MUsT).
  2. Subject has broken, irritated, or unhealed skin.
  3. Subject has an active sunburn.
  4. Subject has used a tanning bed in the previous 4 weeks.
  5. Subject has known skin or autoimmune disease(s).
  6. Subject is anemic or has any chronic condition(s) that may impact blood sample collection.
  7. Women who are pregnant, breastfeeding, or planning to become pregnant during the study or during the 30 days after study drug administration. All female subjects will undergo a serum pregnancy test at Screening, on Day -1, and before discharge from the CRU.
  8. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study.
  9. Subject has known or suspected allergies or sensitivities to any components of the sunscreen formulation.
  10. Subject has clinical laboratory test results (hematology and serum chemistry) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
  11. Subject has used alcohol-, caffeine-, or xanthine-containing products, Seville oranges (sour), grapefruit, or grapefruit juice, within 72 hours before first study drug application.
  12. Subject has a positive test result at Screening for HIV type 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
  13. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
  14. Subject has used any product(s) containing bis-ethylhexyloxyphenol methoxyphenyl triazine (BEMT), such as sunscreen products, hand or body moisturizing lotion, makeup or foundation, hair care product, lip balm, or lipstick within 14 days before Check in (Day -1) and at any time before End-of-Study procedures.
  15. Subject is unable or unwilling to tolerate the scent of sunscreen and the body coverage with sunscreen (i.e., oily appearance and sensation of sunscreen) for the duration of the treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Plasma PK assessment under MUsT Conditions | On the morning of Days 1 through 4, subjects will receive a topical application of the study drug between 07:00 and 10:00 hours followed by 3 more applications each day at 2, 4, and 6 hours after the first application, resulting in study drug application
  • To explore whether the active component, bemotrizinol (BEMT), is absorbed from a high-penetrating sunscreen formulation into the systemic circulation when applied under maximal-use conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC; Rolf Schultz, PhD, Study Director — DSM Nutritional Products, LLC
Locations (1):
- Spaulding Clinical Research LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No